CLINICAL TRIAL: NCT03216824
Title: CVAD-Associated Skin Impairment: A Pilot Study Comparing Dressing to No-Dressing in Adult Allogeneic Stem Cell Transplant Recipients
Brief Title: CVAD-Associated Skin Impairment in Allogeneic Stem Cell Transplant Recipients: Dressing vs No-Dressing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Wendy Hall, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H17-01002
Record Dates: First submitted 2017-05-31; First posted 2017-07-13 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Central Line Complication
MeSH Terms: interventions — Bandages

STUDY DESIGN:
Intervention Model Description: One group will maintain a dressing on the CVAD exit site as per institutional practice. The second group will not cover the CVAD exit site with a dressing (i.e. no-dressing).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dressing (Active Comparator): A dressing is maintained on the CVAD exit site.
  Interventions: Other: Dressing
- No-Dressing (Experimental): The CVAD exit site is not covered with a dressing.
  Interventions: Other: No-Dressing

INTERVENTIONS:
Other: Dressing — A dressing is maintained on the CVAD exit site.
  Arms: Dressing
Other: No-Dressing — The CVAD exit site is not covered with a dressing.
  Arms: No-Dressing

SUMMARY:
Central venous access device (CVAD)-associated skin impairment (CASI) is a common problem in allogeneic hematopoietic stem cell transplant (HSCT) recipients. In this prospective randomized pilot study, dressing the CVAD exit site will be compared to no-dressing with respect to CASI and CVAD-related bloodstream infection (CRBSI) rates in adult outpatient HSCT recipients. The purpose of this study is to gain information that can be used to design a large randomized controlled trial (RCT).

DETAILED DESCRIPTION:
Central venous access device (CVAD)-associated skin impairment (CASI) is common in adult allogeneic hematopoietic stem cell (HSCT) recipients. CASI is defined as chemical, mechanical or microbiological damage to the skin occurring within a 7 cm radius of a CVAD exit site. CASI is associated with discomfort, complex dressing changes, and increased infection risk due to disruption of skin barrier function. Allogeneic hematopoietic stem cell transplant (HSCT) recipients receiving post-transplant care in the outpatient HSCT setting may be at higher risk of CASI. No-dressing of embedded tunneled CVAD (T-CVAD) exit sites may decrease CASI without increased risk of CVAD-related bloodstream infection (CRBSI), but no studies have been conducted to test this hypothesis. A pilot study will determine the practicality of testing this hypothesis. The proposed pilot study will be conducted at an outpatient HSCT clinic located at a large tertiary hospital. The primary aim is to evaluate the logistics of comparing no-dressing to dressing in the outpatient adult allogeneic HSCT population. A total of 26 allogeneic HSCT recipients will be enrolled. Enrollment will commence once the following conditions are met: REB approval, institutional approval, and assignment of an NCT ID number. Eligible participants will have embedded T-CVADs, be within 35 to 60 days of transplant, meet criteria for neutrophil engraftment, and be without pre-existing severe CASI. Participants will be randomized to either a dressing or no-dressing group. A modified version of the Eastern Cooperative Oncology Group (ECOG) skin toxicity scale will be used to grade CASI at baseline and weekly for up to six weeks. Primary and secondary endpoints will be tested statistically to generate estimates of effect size and standard deviations, for the purpose of future study design. Information useful for planning large-scale studies will be reported, such as enrollment metrics, participant compliance, procedure fidelity, and missing data characteristics. Feedback will be collected from participants regarding their study experience.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* 19 years of age or over
* Recipient of an allogeneic HSCT (sibling, haploidentical, or unrelated donor) within the past 35-60 days
* Receiving post-allogeneic HSCT follow-up care at the outpatient HSCT clinic at the study centre
* Possessing a tunneled CVAD with cuff (either Hickman™, Leonard™ or Broviac™) inserted greater than 40 days prior to screening visit
* An embedded T-CVAD exit site (i.e. subcutaneous tissue attached to the internal cuff and prior removal of the exit site suture)
* Documented neutrophil engraftment
* Free of temperature equal to or greater than to 38° C in the past seven days

Exclusion Criteria:

* An infection requiring systemic IV therapy within the last seven days
* A history of abdominal abscess or endocarditis
* Active discharge and/or bleeding from the T-CVAD exit site
* Severe CASI (i.e. greater than grade 3 as per the Modified ECOG Skin Toxicity Scale)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2018-11-04 (Actual); Study Completion 2018-11-04 (Actual)

PRIMARY OUTCOMES:
CVAD-associated skin impairment (CASI) rate | The first CASI assessment will occur within one week of randomization. CASI assessments will be conducted every seven days with up to six assessments in total (i.e. the study follow-up period is six weeks).
  CASI is defined as: chemical, mechanical or microbiological damage to the skin occurring within a 7 cm radius of a CVAD exit site (i.e. the "CASI boundary area"). Skin damage will be measured using a modified ECOG Skin Toxicity Scale. The scale has five levels of measurement with "0" = no CASI, and "1, 2, 3 and 4" corresponding to increasing levels of CASI severity. A finding of CASI of any severity will be counted as one episode of CASI. The rate of CASI will be reported as total CASI episodes.

SECONDARY OUTCOMES:
CVAD-related bloodstream infection (CRBSI) rate | All episodes of CRBSI will be captured during the six week study follow-up period.
  CRBSI is defined as a bloodstream infection linked to a CVAD using a laboratory method with high sensitivity and specificity. In this study differential time to positivity (DTP) will be used to confirm CRBSI. Concomitant peripheral and CVAD blood cultures will be drawn at the new onset of a temperature equal to or greater than 38° C. A set of cultures in which the CVAD culture turns positive two or more hours before a positive peripheral culture will be considered one episode of CRBSI. The rate of CRBSI will be reported according to the number of CRBSI episodes per 1,000 catheter days.
Rate of moderate and severe CVAD-associated skin impairment (CASI) | The first CASI assessment will occur within one week of randomization. CASI assessments will be conducted every seven days with up to six assessments in total.
  All episodes of CASI that meet the modified ECOG Skin Toxicity Scale criteria for levels 2, 3 or 4 will be included to calculate the rate of "moderate and severe" CASI.

OTHER OUTCOMES:
Feasibility Outcome 1: Enrollment rate | Enrollment data will be collected from the start date of enrollment until the date that the total number of required participants has been enrolled. The planned time period is 16 weeks.
  The enrollment rate will be determined by calculating the ratio of participants enrolled to the number of potentially eligible prospective participants invited to participate. The ratio will be reported as a percentage. It will be considered a feasibility concern if > 30% of potentially eligible prospective participants are not enrolled in the study.
Feasibility Outcome 2: Time to complete enrollment | Enrollment data will be collected from the start date of enrollment until the date 26th participant is enrolled. The planned time period is 16 weeks.
  The number of days from the start of enrollment to the end of enrollment (i.e. date 26th participant enrolled) will be calculated. An enrollment period that is > 25% longer than 16 weeks is considered a feasibility concern.
Feasibility Outcome 3: CASI assessment completion rate | CASI assessment data will be collected from the start of enrollment until the date of the final CASI assessment for the last participant enrolled in the study. The planned time period is 22 weeks.
  The CASI assessment completion rate will be determined by calculating the ratio of completed CASI Assessment Forms to required CASI assessments. The CASI Assessment Form includes a 1:1 scale diagram of the CASI boundary area, a key that can be used to indicate specific type(s) of skin impairment on the diagram, and the modified ECOG Skin Toxicity Scale. The CASI assessment completion rate will be expressed as a percentage. A completion rate < 95% is considered a feasibility concern.
Feasibility Outcome 4: Reasons for lack of compliance with CASI assessment | CASI assessment data will be collected from the start of enrollment until the date of the final CASI assessment for the last participant enrolled in the study. The planned time period is 22 weeks.
  The reasons for not completing the CASI Assessment Form will be categorized as: (1) error; (2) participant refused; (3) lack of nurse/researcher time; (4) lack of participant time; (5) participant absent; and (6) other. The frequency of each reason will be reported. A feasibility threshold has not been established for this outcome.
Feasibility Outcome 5: Total number of duplicate CASI assessments | CASI assessment data will be collected from the start of enrollment until the date of the final CASI assessment for the last participant enrolled in the study. The planned time period is 22 weeks.
  A duplicate CASI assessment is scheduled to occur with every fifth CASI assessment in order to assess whether or not consistent data is captured using the CASI Assessment Form. It is possible some scheduled duplicate assessments may not occur. The intention of this outcome is to determine the number of duplicate CASI assessments performed. A feasibility threshold has not been established for this outcome.
Feasibility Outcome 6: Rate of discordant findings for duplicate CASI assessments | CASI assessment data will be collected from the start of enrollment until the date of the final CASI assessment for the last participant enrolled in the study. The planned time period is 22 weeks.
  The ratio of total discordant findings in general to total findings in general with respect to the duplicate CASI Assessment Forms completed will be calculated and expressed as a percentage. If it is found that the discordant findings rate is > 10% this will be considered a feasibility concern (i.e. revision and further testing of the CASI Assessment Form is needed).
Feasibility Outcome 7: Rate of discordant findings for individual elements for duplicate CASI assessments | CASI assessment data will be collected from the start of enrollment until the date of the final CASI assessment for the last participant enrolled in the study. The planned time period is 22 weeks.
  The ratio of discordant findings to total findings for each element of the CASI Assessment Form will be calculated and expressed as a percentage. If it is found that the discordant findings rate is > 10% for a specific element of the CASI Assessment Form, then this will be considered a feasibility concern (i.e. revision and further testing of this specific element in the CASI Assessment Form is needed).
Feasibility Outcome 8: Missing data rate | Data will be collected from the date start of enrollment until the date of the final CASI assessment for the last participant enrolled in the study. The planned time period is 22 weeks.
  The missing data rate will be determined by calculating the ratio of missing data values to total possible data items. The result will be expressed as a percentage. Missing data > 10% is considered a serious feasibility issue.
Feasibility Outcome 9: Type of missing data | Data will be collected from the date start of enrollment until the date of the final CASI assessment for the last participant enrolled in the study. The planned time period is 22 weeks.
  Specific data items with a missing data rate > 5% will be identified. A feasibility threshold has not been established for this outcome.
Feasibility Outcome 10: Participant-dependent compliance | The "Participant Feedback Survey" is completed once. The time point is the last study visit. Survey collection will occur over a planned time period of 16 weeks.
  Participants will be asked to complete a "Participant Feedback Survey" to assess their degree of compliance with study procedures. The survey includes four questions answered using a Likert scale (1-5). Mean scores will be calculated for each question. Mean scores which indicates a feasibility concern have been established a priori for each question.
Feasibility Outcome 11: Duration of Follow-Up | Data will be collected from the start of enrollment until the final visit of the last participant enrolled in the study. The planned time period is 22 weeks.
  If > 20% of participants are withdrawn from the study prior to week six, then this will be considered a significant feasibility issue.
Feasibility Outcome 12: Reasons for Early Withdrawal | Data will be collected from the start of enrollment until the final visit of the last participant enrolled in the study. The planned time period is 22 weeks.
  The reasons for early withdrawal will be reported by frequency according to the following categories: cuff extrusion; absolute neutrophil count < 0.5 x 10^9/L for > 7 consecutive days; temperature greater than or equal to 38 degrees Celsius at one or more time points for > 3 consecutive days; CVAD removed due to positive blood cultures or no longer needed; admission to hospital for a period > 14 days; participant withdrawal from the study. A feasibility threshold has not been established for this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy A. Hall, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers.

REFERENCES:
- [Background] Benhamou E, Fessard E, Com-Nougue C, Beaussier PS, Nitenberg G, Tancrede C, Dodeman S, Hartmann O. Less frequent catheter dressing changes decrease local cutaneous toxicity of high-dose chemotherapy in children, without increasing the rate of catheter-related infections: results of a randomised trial. Bone Marrow Transplant. 2002 Apr;29(8):653-8. doi: 10.1038/sj.bmt.1703511. PMID 12180109
- [Background] Broadhurst D, Moureau N, Ullman AJ; World Congress of Vascular Access (WoCoVA) Skin Impairment Management Advisory Panel. Management of Central Venous Access Device-Associated Skin Impairment: An Evidence-Based Algorithm. J Wound Ostomy Continence Nurs. 2017 May/Jun;44(3):211-220. doi: 10.1097/WON.0000000000000322. PMID 28353488
- [Background] Dix CH, Yeung DT, Rule ML, Ma DD. Essential, but at what risk? A prospective study on central venous access in patients with haematological malignancies. Intern Med J. 2012 Aug;42(8):901-6. doi: 10.1111/j.1445-5994.2011.02596.x. PMID 21981058
- [Background] Gillies D, O'Riordan E, Carr D, O'Brien I, Frost J, Gunning R. Central venous catheter dressings: a systematic review. J Adv Nurs. 2003 Dec;44(6):623-32. doi: 10.1046/j.0309-2402.2003.02852.x. PMID 14651685
- [Background] Keeler M. Central line practice in Canadian blood and marrow transplant. Can Oncol Nurs J. 2014 Spring;24(2):67-77. doi: 10.5737/1181912x2426771. English, French. PMID 24902424
- [Background] Keeler, M., Haas, B., Northam, S., Nieswiadomy, M., McConnel, C., & Savoie, L. Analysis of costs and benefits of transparent, gauze, or no dressing for a tunnelled central venous catheter in Canadian stem cell transplant recipients. Canadian Oncology Nursing Journal. 25(3): 289-298, 2015.
- [Background] Lawrence JA, Seiler S, Wilson B, Harwood L. Shower and no-dressing technique for tunneled central venous hemodialysis catheters: a quality improvement initiative. Nephrol Nurs J. 2014 Jan-Feb;41(1):67-72; quiz 73. PMID 24689266
- [Background] Mimoz O, Lucet JC, Kerforne T, Pascal J, Souweine B, Goudet V, Mercat A, Bouadma L, Lasocki S, Alfandari S, Friggeri A, Wallet F, Allou N, Ruckly S, Balayn D, Lepape A, Timsit JF; CLEAN trial investigators. Skin antisepsis with chlorhexidine-alcohol versus povidone iodine-alcohol, with and without skin scrubbing, for prevention of intravascular-catheter-related infection (CLEAN): an open-label, multicentre, randomised, controlled, two-by-two factorial trial. Lancet. 2015 Nov 21;386(10008):2069-2077. doi: 10.1016/S0140-6736(15)00244-5. Epub 2015 Sep 18. PMID 26388532
- [Background] Nagai T, Kohsaka S, Anzai T, Yoshikawa T, Fukuda K, Sato T. Low incidence of catheter-related complications in patients with advanced pulmonary arterial hypertension undergoing continuous epoprostenol infusion. Chest. 2012 Jan;141(1):272-273. doi: 10.1378/chest.11-1893. No abstract available. PMID 22215838
- [Background] O'Grady NP, Alexander M, Burns LA, Dellinger EP, Garland J, Heard SO, Lipsett PA, Masur H, Mermel LA, Pearson ML, Raad II, Randolph AG, Rupp ME, Saint S; Healthcare Infection Control Practices Advisory Committee (HICPAC). Guidelines for the prevention of intravascular catheter-related infections. Clin Infect Dis. 2011 May;52(9):e162-93. doi: 10.1093/cid/cir257. Epub 2011 Apr 1. No abstract available. PMID 21460264
- [Background] Olson K, Rennie RP, Hanson J, Ryan M, Gilpin J, Falsetti M, Heffner T, Gaudet S. Evaluation of a no-dressing intervention for tunneled central venous catheter exit sites. J Infus Nurs. 2004 Jan-Feb;27(1):37-44. doi: 10.1097/00129804-200401000-00006. PMID 14734986
- [Background] Orsino, L., Bargelli, A., Cappucciati, L., Fanchin, G., Galati, G., Manzin, F., ... Vendemiati, S. Observational study of SorbaView® 2000, SorbaView® ultimate and SecureView® port AFZ dressings used on central venous catheters in eleven italian oncology, hematology and pain centers. Journal of the Association for Vascular Access, 14(1): 14-19, 2009.
- [Background] Petrosino B, Becker H, Christian B. Infection rates in central venous catheter dressings. Oncol Nurs Forum. 1988 Nov-Dec;15(6):709-17. No abstract available. PMID 3144709
- [Background] Laura R, Degl'Innocenti M, Mocali M, Alberani F, Boschi S, Giraudi A, Arnaud MT, Zucchinali R, Paris MG, Dallara R, Thaler S, Perobelli G, Parfazi S, De Lazzer T, Peron G. Comparison of two different time interval protocols for central venous catheter dressing in bone marrow transplant patients: results of a randomized, multicenter study. The Italian Nurse Bone Marrow Transplant Group (GITMO). Haematologica. 2000 Mar;85(3):275-9. PMID 10702816
- [Background] Renaud B, Brun-Buisson C; ICU-Bacteremia Study Group. Outcomes of primary and catheter-related bacteremia. A cohort and case-control study in critically ill patients. Am J Respir Crit Care Med. 2001 Jun;163(7):1584-90. doi: 10.1164/ajrccm.163.7.9912080. PMID 11401878
- [Background] Rosenthal VD, Guzman S, Migone O, Crnich CJ. The attributable cost, length of hospital stay, and mortality of central line-associated bloodstream infection in intensive care departments in Argentina: A prospective, matched analysis. Am J Infect Control. 2003 Dec;31(8):475-80. doi: 10.1016/j.ajic.2003.03.002. PMID 14647110
- [Background] Safdar N, Fine JP, Maki DG. Meta-analysis: methods for diagnosing intravascular device-related bloodstream infection. Ann Intern Med. 2005 Mar 15;142(6):451-66. doi: 10.7326/0003-4819-142-6-200503150-00011. PMID 15767623
- [Background] Shivnan JC, McGuire D, Freedman S, Sharkazy E, Bosserman G, Larson E, Grouleff P. A comparison of transparent adherent and dry sterile gauze dressings for long-term central catheters in patients undergoing bone marrow transplant. Oncol Nurs Forum. 1991 Nov-Dec;18(8):1349-56. PMID 1762975
- [Background] Silveira RC, Braga FT, Garbin LM, Galvao CM. The use of polyurethane transparent film in indwelling central venous catheter. Rev Lat Am Enfermagem. 2010 Nov-Dec;18(6):1212-20. doi: 10.1590/s0104-11692010000600023. PMID 21340288
- [Background] Timsit JF, Schwebel C, Bouadma L, Geffroy A, Garrouste-Orgeas M, Pease S, Herault MC, Haouache H, Calvino-Gunther S, Gestin B, Armand-Lefevre L, Leflon V, Chaplain C, Benali A, Francais A, Adrie C, Zahar JR, Thuong M, Arrault X, Croize J, Lucet JC; Dressing Study Group. Chlorhexidine-impregnated sponges and less frequent dressing changes for prevention of catheter-related infections in critically ill adults: a randomized controlled trial. JAMA. 2009 Mar 25;301(12):1231-41. doi: 10.1001/jama.2009.376. PMID 19318651